CLINICAL TRIAL: NCT05155358
Title: Study on the Establishment of a System for Early Warning and Prognostic Evaluation of Patients With Heat Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212173
Record Dates: First submitted 2021-12-08; First posted 2021-12-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Heat Stroke; Early Waking; MODS; Proteinosis; Liver Injury; Kidney Injury
MeSH Terms: conditions — Heat Stroke; Sleep Initiation and Maintenance Disorders; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, PBMC, plasma exosome miRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control group: Healthy volunteers
  Interventions: Diagnostic Test: Peripheral blood test
- Patients within the acute phase of disease: Patients within 24 hours after onset
  Interventions: Diagnostic Test: Peripheral blood test
- Recovery stage of disease: Organ dysfunction was corrected, The patient had no obvious discomfort.
  Interventions: Diagnostic Test: Peripheral blood test

INTERVENTIONS:
Diagnostic Test: Peripheral blood test — Collect peripheral blood to separate and extract plasma, PBMC, and plasma exosomal miRNA, and sequence to find indicators related to disease deterioration and prognosis

SUMMARY:
Heat stroke is a clinical syndrome with high incidence and high fatality rate in summer. Patients with liver, kidney, and brain damage are prone to secondary MODS, and the prognosis is poor due to high medical costs. At present, there is no unified diagnostic criteria for acute liver injury associated with heat stroke, and the commonly used prognosis scores are rarely included in liver injury indicators, which is not good for practicality.

DETAILED DESCRIPTION:
The project intends to collect the peripheral blood of the normal population, the 24 hours after the onset of heat stroke and the patients in the recovery period, to separate and extract plasma, PBMC, and plasma exosomal miRNA, and sequence to search for indicators related to disease deterioration and prognosis, construct and verify the early warning and prognosis evaluation system of the disease.

On this basis, the researcher explore cellular and molecular mediated pathological mechanisms of heat stroke, and then clarify the treatment target of heat stroke.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily signs an informed consent form;
2. Adult patients who meet the criteria for heat stroke;
3. Heat stroke is defined as heat stroke (Heat Stroke, HS) is a serious fatal disease caused by heat injury factors acting on the body, accompanied by multiple organ damage.

Exclusion Criteria:

1. Age <18 years old or >90 years old;
2. Patients with advanced tumors, Pregnancy or lactation;
3. Patients who missed out during treatment and whose data are incomplete.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy Volunteers with routine physical examination;
  2. Heat stroke is defined as heat stroke (Heat Stroke, HS) is a serious fatal disease caused by heat injury factors acting on the body, accompanied by multiple organ(liver,kindey, lung ect) dysfunction.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis | Day 30 and Day 90
  Rate of Surviving or Died Participants with Heat Stroke

SECONDARY OUTCOMES:
Heat Stroke-associated kindey injury | Day 0, Day 7 and On the day of discharge after improvement
  Concentration of Creatinine(Cr)>2 mg/dl or Urine output < 500ml/Day
Heat Stroke-associated liver injury | Day 0, Day 7 and On the day of discharge after improvement
  Concentration of ALT or AST >80 U/L, Concentration of TBIL>2mg/dl（34μmol/l）

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Jia, Study Chair — The First Affillated Hospital,the Air Force Medical University
Locations (1):
- The First Affillated Hospital,the Air Force Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No